CLINICAL TRIAL: NCT07073261
Title: PROspective Multiethnic Validation of the BEhçet's Syndrome Overall Damage Index (BODI): the PROBE Study
Brief Title: Prospective Multiethnic Validation of the Behçet's Syndrome Overall Damage Index (BODI)
Acronym: PROBE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: Hôpital de Hautepierre (Other); University of Siena (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (IDIBAPS), Universitat de Barcelona, Barcelona, Spain. (Unknown); Università degli Studi di Ferrara (Other); Tabriz University of Medical Sciences (Other); University of Bari (Other); Cairo University (Other); Tehran University of Medical Sciences (Other); Ibn Sina University Hospital, Rabat, Morocco (Other); Istanbul University (Other); Nazarbayev University School of Medicine (Unknown); Aristotle University Of Thessaloniki (Other); Mayo Clinic (Other); Centro Hospitalar do Porto (Other); Centro Hospitalar do Tâmega e Sousa (Other); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Matteo Piga, Associate Professor of Rheumatology, University of Cagliari
Other Study IDs: PROBE
Record Dates: First submitted 2025-06-27; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Behçet's Syndrome (BS)
Keywords: PROBE; Behçet's syndrome; Damage; Behçet's syndrome Overall Damage Index; BODI; Geographic variability; Damage accrual; Hospitalization; Mortality
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PROBE is an observational multicenter cohort study, consisting of a cross-sectional and a 5-years prospective phase, designed to target the major study objectives, such as testing the comprehensiveness of the Behçet's syndrome Overall Damage Index (BODI) in a wide and ethnically heterogeneous cohort of Behçet's syndrome patients, and investigating how damage assessed by the BODI correlates with other major long-term disease outcomes (5-years mortality and hospitalization rates).

DETAILED DESCRIPTION:
Behçet's syndrome (BS) is a multisystem inflammatory disease of unknown etiology, characterized by strong genetic background, distinctive geographic distribution, and wide variability in clinical presentation. Disease activity related to BS as well as chronic exposure to medications may lead to the development and accrual of irreversible organ damage resulting in impairment of quality of life, disability, and increased mortality. For these reasons, organ damage was included in the Outcome Measures in Rheumatology (OMERACT) outcome core set for BS. The Behçet's syndrome Overall Damage Index (BODI) is a recently developed tool to identify and measure organ damage in BS. The BODI is grounded in a solid evidence-based and consensus-based methodology, and its preliminary validation on a multicenter cohort of Southern European patients showed highly promising performance in terms of comprehensiveness, specificity, reliability, sensitivity to change, and feasibility. Nevertheless, a prospective validation with a wider and ethnically heterogeneous cohort of BS patients is needed to generally evaluate the impact of those BODI items seldom recorded or absent in the preliminary validation cohort and to weigh the damage items depending on their relevance for predicting major outcomes.

PROBE is an observational multicenter cohort study, consisting of a cross-sectional and a 5-years prospective phase, designed to target the major study objectives, such as testing the comprehensiveness of the BODI (content validity) in a wide and ethnically heterogeneous cohort of BS patients, and investigating how damage assessed by the BODI correlates with other major long-term disease outcomes (criterion validity), with the ultimate goal of drafting a weighing system for each BODI item. Specific objectives are reported as follow:

1. To test the comprehensiveness of the instrument in a wide and ethnically heterogeneous cohort of BS patients, evaluating the prevalence of those BODI items seldom recorded or absent in the preliminary validation cohort.
2. To describe possible differences in the entity and type of damage accrual in BS patients from different geographical areas.
3. To identify the factors independently associated with damage development and accrual.
4. To investigate the association between the results of the baseline BODI measurement (BODI ≥1, BODI score, and BODI ranking) and the 5-years mortality rate.
5. To investigate the association between the results of the baseline BODI measurement (BODI ≥1, BODI score, and BODI ranking)and the 5-years hospitalization rate.
6. To weigh each item of damage depending on their relevance in predicting mortality.

The study population will consist of consecutive BS patients diagnosed according to the International Criteria for Behçet's Disease (ICBD) or International Study Group (ISG) classification criteria, recruited in Centers with expertise for BS. Demographic and clinical data will be collected at the time of recruitment (baseline, T0) and then annually (± 1 month) for 5 years. Overall, 6 visits are planned to be recorded (T0, T1, T2, T3, T4, T5).

During the study, patients will undergo a routine clinical assessment, as scheduled in their followup program. No further clinical, laboratory or instrumental investigations are required in addition to those provided according to good clinical practice. Treatment prescription will be evaluated by each investigator independently from the study and according to the international and local guidelines and the good clinical practice.

Descriptive statistics will be performed to report on the prevalence and amount of damage, as assessed by the BODI. In the whole study cohort and different geographical sub-groups, the damage will be described as:

* prevalence of any damage (BODI ≥1);
* prevalence of any damage in the different BODI domains;
* mean (SD) or median (IQR) BODI score.

Ranking of the BODI score will be developed, using a multistate model, depending on the distribution of damage in the whole population.

Univariate and multivariate regression models will be implemented to investigate the significant difference between ethnic/geographic groups in terms of prevalence and amount of damage accrual. Similarly, univariate and multivariate regression models will be implemented to investigate independent factors associated with the development or accrual of damage, as assessed by the BODI. Multivariate Cox proportional hazards regression models will be created to assess the effect of damage (BODI score, BODI ≥1, BODI ranking) on subsequent risk of death with adjustment for covariates, including gender, age, disease duration at enrollment, history of major organ involvement, disease activity at enrolment, comorbidities (onset before BS diagnosis). Results will be presented as hazard ratios with their corresponding 95% confidence intervals. Statistical significance will be defined as a P-value <0.05. Finally, adjusted survival estimates obtained from these Cox regression models were plotted as survival curves.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BS according to ICBD or ISG criteria.

Exclusion Criteria:

* Subjects unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow interval visits.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of consecutive Behçet's syndrome (BS) patients, coming from 11 different countries, diagnosed according to the ICBD or ISG classification criteria, recruited in Centers with expertise for BS.
Sampling Method: Non-Probability Sample
Enrollment: 970 (Actual)
Dates: Start 2021-07-23 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
5-years mortality rate | 5 years
  Correlation between the irreversible organ damage measured by the BEhçet's syndrome Overall Damage Index (BODI) and the 5-years mortality rate.
5-years hospitalization rate | 5 years
  Correlation between the irreversible organ damage measured by the BEhçet's syndrome Overall Damage Index (BODI) and the 5-years hospitalization rate.

SECONDARY OUTCOMES:
Organ damage accrual measured by the BEhçet's syndrome Overall Damage Index (BODI) | 5 years
  Annual rate of increase in irreversible organ damage measured by the BEhçet's syndrome Overall Damage Index (BODI).
Differences in annual rate of increase in organ damage in patients coming from different geographical areas. | 5 years
  Differences in annual rate of increase in organ damage measured by the BEhçet's syndrome Overall Damage Index (BODI) in patients coming from different geographical areas, categorized in:
  * Europe
  * Middle East
  * North Africa
  * Americas
  * Central Asia

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Piga, Medicine and Surgery, Principal Investigator — University of Cagliari
Locations (1):
- Rheumatology Unit, University and AOU of Cagliari, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT07073261/Prot_000.pdf